CLINICAL TRIAL: NCT01572532
Title: Maternal Genitourinary Infections and Adverse Perinatal Outcomes in Sylhet District, Bangladesh
Brief Title: Maternal Genitourinary Infections and Adverse Perinatal Outcomes
Acronym: MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003063; 1R01HD066156-01 (NIH)
Record Dates: First submitted 2011-12-15; First posted 2012-04-06 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Maternal Infection Affecting Newborn
Keywords: Adverse Perinatal Outcomes; Treatment of abnormal vaginal flora
MeSH Terms: interventions — Referral and Consultation; Mass Screening

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Screening and Treatment (Experimental): CHWs will collect urine and vaginal samples for all women enrolled. In the control clusters, every eighth woman enrolled will receive the screening-treatment protocol in order to determine the baseline prevalence of these infections in the control areas for comparison. Vaginal specimens will be collected via sterile self-administered vaginal swabs. The women will be instructed by the CHW to insert a Dacron swab ~4-5 cm into the vagina, allow the swab to stand for 15 seconds, and then rotate 360 degrees prior to withdrawal. The CHW will gently roll out the swab onto a plain glass slide and allow to air dry prior to transport to Sylhet field laboratory.
  A midstream urine specimen will be obtained for urine culture. The mother will be instructed to separate the labia and collect 20-30mL of midstream urine into a sterile container which will be immediately refrigerated in a cool specimen box.
  Interventions: Other: Screening treatment and referral
- Control Arm (No Intervention): Standard care will be administered, including antenatal and postnatal care. In the control clusters, every eighth woman enrolled will receive the screening-treatment protocol in order to determine the baseline prevalence of these infections in the control areas for comparison.

INTERVENTIONS:
Other: Screening treatment and referral — Women who are symptomatic at any study visit will be immediately referred to the sub-district hospital for full evaluation and treatment and will be visited on the following day to follow clinical status and ensure referral compliance. Referral will be reinforced by arranging transportation to the sub-district hospital and payment of hospital fees if the family is unable to afford out-of-pocket expenses. CHWs will conduct a home visit to women with positive test results within 24 hours of receiving the results to initiate treatment. All asymptomatic women will be treated for positive test results. For symptomatic women, the CHW will confirm the woman's clinical and treatment status, and provide treatment to those women who have not already received the appropriate treatment at the sub-district hospital for their infection.
  Antibiotic Treatment Regimens AVF: Oral clindamycin 300 mg per oral (po) twice daily (bid) for 5 days.UTI: Macrobid/Nitrofurantoin 100 mg po bid x 7 days.
  Other Names: Screening and Treatment of Abnormal Vaginal Flora; Screening and Treatment of Urinary Tract Infections
  Arms: Intervention Screening and Treatment

SUMMARY:
The primary aim of this study is to determine the impact of community-based screening and treatment of abnormal vaginal flora and urinary tract infections in early pregnancy (13-19 weeks) on preterm live birth in Sylhet district, Bangladesh.

Hypothesis 1: Community-based screening and treatment of abnormal vaginal flora (Nugent score >4) and urinary tract infections in early pregnancy (13-19 weeks) will reduce the population rate of preterm live birth by at least 15%.

The secondary aims of this study are:

* To determine the impact of community-based screening and treatment of abnormal vaginal flora and urinary tract infections on the:

  * proportion of pregnancies with outcomes occurring prior to 37 weeks (late miscarriage, preterm still birth and preterm live birth); and
  * proportion of babies with early onset neonatal sepsis.
* To determine the prevalence of abnormal vaginal flora and urinary tract infections, including asymptomatic bactiuria, among pregnant women in Sylhet district, Bangladesh.
* To evaluate the accuracy of simple, low-cost, point of care diagnostic tests for detecting bacterial vaginosis and urinary tract infections by community health workers in a rural, developing country setting.

DETAILED DESCRIPTION:
Burden of Maternal Genitourinary Tract Infections: Genital and urinary tract (GU) infections may be due to endogenous or sexually transmitted pathogens, and are estimated to affect up to 41% of women of reproductive age globally, although there is wide regional, country, and population specific variation (Table 1). These estimates, however, may underestimate the burden in developing countries, as 60-80% of GU infections are asymptomatic in pregnant women [1], and furthermore many women never receive appropriate medical care in resource poor settings.

Several epidemiologic studies have been conducted in Bangladesh reporting the prevalence of GU infections in different populations [2-15]. Genital tract infections, particularly sexually transmitted infections are common among urban and high risk populations, i.e. commercial sex workers. In rural Bangladesh, the burden of diseases associated with bacterial vaginosis (BV) (5.9-18.9%) [3, 4] and asymptomatic bactiuria (12%) are high [12]. In urban areas, mostly Dhaka, the prevalence of BV is higher; one study reported a prevalence of 28% [8]. There is no known data on the prevalence of intermediate vaginal flora in Bangladesh. The prevalence of sexually transmitted infections including Gonorrhea, Chlamydia, Trichomonas and Syphilis are high among high risk urban populations of Bangladesh but generally low in rural areas. Given these prevalence data, we postulate that among pregnant women of rural Sylhet district in Bangladesh, BV and UTI are the most prevalent GU infections.

Rationale for screening and treating asymptomatic women The rationale for treating asymptomatic bacterial vaginosis (Nugent score 7-10) and asymptomatic intermediate flora (Nugent score 4-6) is based on data: 1) showing their association with adverse pregnancy outcomes[38], and 2) several promising trials showing that treatment may reduce preterm birth[39, 40]. Up to 84% of bacterial vaginosis cases are asymptomatic [23]. In a meta-analysis of 32 studies in developed and developing countries by Leitich et al, asymptomatic BV (Nugent score 7-10) was associated with a 6.32 times elevated risk of late miscarriage (95% CI 3.65-10.94) and 2.16 times (95% CI 1.56-3.00) increased risk of preterm birth. The association with preterm birth was higher when BV was detected in early pregnancy (<16 weeks, OR 2.97, 95% CI 1.48-5.98)[38]. Among women with a prior history of preterm birth, Hauth and colleagues found that screening and treatment of asymptomatic BV (Nugent score 7-10) with metronidazole and erythromycin at 22 weeks gestation significantly reduced the incidence of preterm birth from 46% in the placebo group to 31% in the treatment group [41]. In the multi-center NICHD BV trial, 1953 women with asymptomatic BV between 16-24 weeks of gestation were randomized to receive two doses of metronidazole (2g) or placebo; however, treatment did not significantly affect preterm delivery or other adverse perinatal outcomes [42].

Intermediate vaginal flora (Nugent score 4-6) is a heterogeneous condition which has been also associated with elevated risk of preterm birth and neonatal infections [43-46]. Intermediate vaginal flora comprises 15% of all abnormal vaginal flora (Nugent score >=4) [39]. In a recent trial, Ugwumadu et al reported that early (12-22 weeks of gestation) screening and treatment for abnormal vaginal flora (Nugent score >4) with 5 days of oral clindamycin resulted in a significant reduction in spontaneous preterm birth rate (12% in placebo vs. 5% in treatment group) and late miscarriage (13-24 weeks; 4% in placebo vs. 1% in treatment group) [39]. Similarly, Lamont et al reported that early (13-20 week) treatment of abnormal vaginal flora (Nugent score >4) with intravaginal clindamycin reduced the incidence of preterm birth by 60% [40]. Potential explanations for the treatment effect in the 2 later trials may include: 1) the earlier timing of treatment, prior to the amniotic membranes sealing the uterus at 20 weeks [47], which may thus prevent early ascension of bacteria into the intrauterine cavity; 2) antibiotic choice: 5-7 day course of clindamycin, which has greater activity against Mobiluncus and atypical Mycoplasma species vs. 2 days of metronidazole [26]; and 3) treatment of abnormal vaginal flora in Ugwumadu et al and Lamont et al, vs. treatment of BV only in the NICHD trial. A Cochrane meta-analysis concluded that the risk of preterm birth was significantly reduced by treatment of abnormal vaginal flora (Nugent score >4) (2 trials, 894 women; OR 0.51, 95% CI 0.32-0.81). Thus, in low-resource settings such as in rural Bangladesh, where both BV and preterm birth are prevalent, treatment of abnormal vaginal flora in early pregnancy may hold promise in reducing the incidence of preterm birth, and an evaluation in well-conducted community-based randomized trials is needed.

ELIGIBILITY:
Inclusion Criteria:

All women who become pregnant in the study area will be eligible to participate in the trial. We will identify women with missed periods through monthly surveillance by health workers and identify pregnant women by positive pregnancy test conducted by CHWs. Thus enrollment may begin as soon as 5 weeks gestation and will continue until 19 weeks gestation. A sample of women who are enrolled early in gestation (<12 weeks), will be considered for enrolment in the gestational age sub-study. The first CHW visit for screening for abnormal vaginal flora and urinary tract infection will occur after the initial enrollment between 13-19 weeks. Their infants will enrolled as well.

Exclusion Criteria:

Subjects will be excluded from the study if they have no recall or uncertain report of LMP (due to lactational amenorrhea, recent discontinuation of contraceptive or irregular menses), history of irregular bleeding due to injectable depoprovera, or history of severe chronic disease based on their self-reported history on a medical history checklist. For women reporting a missed period during pregnancy surveillance, the CHW will perform a urine pregnancy test to confirm the pregnancy and keep a log of all positive pregnancy tests and LMP.

Pregnant women who are uncertain or refuse to participate at the initial visit will be allowed time to consider and enroll at the next study visit if they still meet inclusion criteria. Women will be given information regarding the study and CHWs will answer questions for both themselves and the family. If a woman is not certain whether she would like to participate, she will be allowed 1 week to consider participation, and the CHW will return in 1 week to revisit participation and answer any additional questions. If the woman refuses to participate at any visit, she will no longer be approached to participate.

Families can withdraw from the study at any time, and study staff will be available to answer questions families may have at any time.

Ages: 1 Minute to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9712 (Actual)
Dates: Start 2010-08; Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
Number of preterm births reduced by community-based screening and treatment of abnormal vaginal flora and urinary tract infections in early pregnancy (13-19 weeks) | 5 years
  Determine the impact of community-based screening and treatment of abnormal vaginal flora and urinary tract infections in early pregnancy (13-19 weeks) on preterm live birth in Sylhet district, Bangladesh.

SECONDARY OUTCOMES:
Proportion of early outcomes | 5 years
  Proportion of pregnancies with outcomes occurring prior to 37 weeks (late miscarriage, preterm still birth and preterm live birth) in Sylhet, Bangladesh
Proportion of infants with neonatal sepsis | 5 years
  Proportion of babies with early onset neonatal sepsis in Sylhet, Bangladesh
Prevalance abnormal vaginal flora | 5 years
  Prevalence of abnormal vaginal flora and urinary tract infections, including asymptomatic bactiuria, among pregnant women in Sylhet district, Bangladesh
Accuracy of diagnostic tests for detecting bacterial vaginosis | 5 years
  Accuracy of simple, low-cost, point of care diagnostic tests for detecting bacterial vaginosis and urinary tract infections by community health workers in a rural, developing country setting (Sylhet, Bangladesh)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah H Baqui, MBBS, MPH, DrPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Community Based, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee AC, Mullany LC, Quaiyum M, Mitra DK, Labrique A, Christian P, Ahmed P, Uddin J, Rafiqullah I, DasGupta S, Rahman M, Koumans EH, Ahmed S, Saha SK, Baqui AH; Projahnmo Study Group in Bangladesh. Effect of population-based antenatal screening and treatment of genitourinary tract infections on birth outcomes in Sylhet, Bangladesh (MIST): a cluster-randomised clinical trial. Lancet Glob Health. 2019 Jan;7(1):e148-e159. doi: 10.1016/S2214-109X(18)30441-8. PMID 30554751
- [Derived] Lee ACC, Whelan R, Bably NN, Schaeffer LE, Rahman S, Ahmed S, Moin SMI, Begum N, Quaiyum MA, Rosner B, Litch JA, Baqui AH, Wylie BJ. Prediction of gestational age with symphysis-fundal height and estimated uterine volume in a pregnancy cohort in Sylhet, Bangladesh. BMJ Open. 2020 Mar 12;10(3):e034942. doi: 10.1136/bmjopen-2019-034942. PMID 32169927
- [Derived] Lee AC, Mullany LC, Ladhani K, Uddin J, Mitra D, Ahmed P, Christian P, Labrique A, DasGupta SK, Lokken RP, Quaiyum M, Baqui AH; Projahnmo Study Group. Validity of Newborn Clinical Assessment to Determine Gestational Age in Bangladesh. Pediatrics. 2016 Jul;138(1):e20153303. doi: 10.1542/peds.2015-3303. Epub 2016 Jun 16. PMID 27313070
- [Derived] Lee AC, Quaiyum MA, Mullany LC, Mitra DK, Labrique A, Ahmed P, Uddin J, Rafiqullah I, DasGupta S, Mahmud A, Koumans EH, Christian P, Saha S, Baqui AH; Projahnmo Study Group. Screening and treatment of maternal genitourinary tract infections in early pregnancy to prevent preterm birth in rural Sylhet, Bangladesh: a cluster randomized trial. BMC Pregnancy Childbirth. 2015 Dec 7;15:326. doi: 10.1186/s12884-015-0724-8. PMID 26643558